CLINICAL TRIAL: NCT05165147
Title: Analysis the Positive Status of Tumor Markers Among Physical Examination Population in a Tertiary Grade A Class Hospital
Brief Title: Analysis the Positive Rate of Tumor Markers Among Physical Examination Population
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006761-M2021321
Record Dates: First submitted 2021-10-20; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-09

CONDITIONS: Tumor
Keywords: physical examination population; tumor marker; TM
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- physical examination population: From January 2019 to December 2019, who underwent physical examination in Peking University Third Hospital were included in the study.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
To analyze the positive rate of tumor markers (TM) among health examination population in a tertiary grade A class hospital, compare the differences between different age and sex groups, and explore the possible influencing factors of TM positive.

DETAILED DESCRIPTION:
From January 2019 to December 2019, who underwent physical examination in Peking University Third Hospital were included in the study. The expression levels of carcinoembryonic antigen (CEA),α-fetoprotein (AFP), carbohydrate antigen 19-9 (CA 19-9), carbohydrate antigen-125 (CA-125), carbohydrate antigen 72-4(CA 72-4), carbohydrate antigen 15-3 (CA 15-3), carbohydrate antigen 242(CA 242), squamous cell carcinoma antigen（SCC）, CYFRA21-1, total prostate-specific antigen (TPSA ) , free prostate-specific antigen(FPSA), neuron specific enolase(NSE) were detected by Electro chemistry luminescence method. The positive rates of TM were analyzed by descriptive statistical method Explore. The differences between different age and sex groups and the influencing factors were explored by statistic by Inferential statistical method.

ELIGIBILITY:
Inclusion Criteria:

* Those who have taken a physical examination and performed at least one TM test

Exclusion Criteria:

* Basic information is missing and cannot be retrieved
* The patient was diagnosed with malignant tumor before examination
* Those who have not done any TM tests

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: rom January 2019 to December 2019, who underwent physical examination in Peking University Third Hospital were included in the study.
Sampling Method: Probability Sample
Enrollment: 26891 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
the positive rate of carcinoembryonic antigen（CEA） | 2019.01.01-2019.12.31
  The proportion of abnormal CEA in physical examination population was calculated. The range of normal value ： CEA≤5 ng/mL.
the positive rate of α-fetoprotein（AFP） | 2019.01.01-2019.12.31
  The proportion of abnormal AFP in physical examination population was calculated. The range of normal value ： AFP≤20 ng/mL.
the positive rate of carbohydrate antigen 19-9（CA 19-9） | 2019.01.01-2019.12.31
  The proportion of abnormal CA 19-9 in physical examination population was calculated. The range of normal value ： CA 19-9≤39 U/mL.
the positive rate of carbohydrate antigen 125（CA 125） | 2019.01.01-2019.12.31
  The proportion of abnormal CA 125 in physical examination population was calculated. The range of normal value ： CA 125≤35 U/mL.
the positive rate of carbohydrate antigen 72-4（CA 72-4） | 2019.01.01-2019.12.31
  The proportion of abnormal CA 72-4 in physical examination population was calculated. The range of normal value ： CA 72-4≤8.2 U/mL.
the positive rate of carbohydrate antigen 15-3（CA 15-3） | 2019.01.01-2019.12.31
  The proportion of abnormal CA 15-3 in physical examination population was calculated. The range of normal value ： CA 15-3≤25 IU/mL.
the positive rate of carbohydrate antigen 242（CA 242） | 2019.01.01-2019.12.31
  The proportion of abnormal CA 242 in physical examination population was calculated. The range of normal value ：CA 242≤20 U/mL.
the positive rate of squamous cell carcinoma antigen（SCC） | 2019.01.01-2019.12.31
  The proportion of abnormal SCC in physical examination population was calculated. The range of normal value ：SCC≤1.5 ng/mL.
the positive rate of Cytokeratin 19 fragment 21-1（CYFRA21-1） | 2019.01.01-2019.12.31
  The proportion of abnormal CYFRA21-1 in physical examination population was calculated. The range of normal value ：CYFRA21-1≤3.3 ng/mL.
the positive rate of total prostate-specific antigen（ TPSA） | 2019.01.01-2019.12.31
  The proportion of abnormal TPSA in physical examination population was calculated. The range of normal value ：TPSA≤4 ng/mL.
the positive rate of free prostate-specific antigen（ FPSA） | 2019.01.01-2019.12.31
  The proportion of abnormal FPSA in physical examination population was calculated. The range of normal value ：FPSA≤1 ng/mL.
the positive rate of neuron specific enolase（ NSE） | 2019.01.01-2019.12.31
  The proportion of abnormal NSE in physical examination population was calculated. The range of normal value ：NSE≤17 ng/mL.

SECONDARY OUTCOMES:
age | 2019.01.01-2019.12.31
  the age of physical examination population.
the measured value of systolic blood pressure (SBP) | 2019.01.01-2019.12.31
  SBP measured on the day of physical examination.Unit of measure：mmHg
the measured value of diastolic blood pressure (DBP) | 2019.01.01-2019.12.31
  DBP measured on the day of physical examination.Unit of measure：mmHg
the measured value of fasting bood glucose (FBG) | 2019.01.01-2019.12.31
  FBG measured on the day of physical examination.Unit of measure：mmol/L
the measured value of total cholesterol (TC) | 2019.01.01-2019.12.31
  TC measured on the day of physical examination.Unit of measure：mmol/L
the measured value of Triglyceride (TG) | 2019.01.01-2019.12.31
  TG measured on the day of physical examination.Unit of measure：mmol/L
the measured value of high density lipoprotein-cholesterol (HDL-C) | 2019.01.01-2019.12.31
  HDL-C measured on the day of physical examination.Unit of measure：mmol/L
the measured value of low density lipoprotein-cholesterol (LDL-C) | 2019.01.01-2019.12.31
  LDL-C measured on the day of physical examination.Unit of measure：mmol/L
the measured value of height | 2019.01.01-2019.12.31
  height measured on the day of physical examination.Unit of measure：cm
the measured value of weight | 2019.01.01-2019.12.31
  height measured on the day of physical examination.Unit of measure：kg
Body Mass Index (BMI) | 2019.01.01-2019.12.31
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, doctorate, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
no share

REFERENCES:
- [Result] Welch HG, Albertsen PC. Reconsidering Prostate Cancer Mortality - The Future of PSA Screening. N Engl J Med. 2020 Apr 16;382(16):1557-1563. doi: 10.1056/NEJMms1914228. No abstract available. PMID 32294352